CLINICAL TRIAL: NCT07230249
Title: Effect of a Behavioral Intervention Delivered Via Telegram Messenger on Smoking Cessation in Patients After Myocardial Infarction: The TELEGRAM-MI Randomized Controlled Trial
Brief Title: Telegram Messenger Support for Smoking Cessation After Heart Attack
Acronym: TELEGRAM-MI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ITMO University (Other)
Responsible Party: Principal Investigator, Mikhail Kuznetsov, Chief Investigator, Cardiologist, ITMO University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TELEGRAM-MI
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Myocardial Infarction (MI); Tobacco Use; Smoking Cessation
Keywords: Telegram; Chatbot; Digital Health; Behavioral Intervention; Secondary Prevention; Randomized Controlled Trial; Cardiac Rehabilitation
MeSH Terms: conditions — Myocardial Infarction; Tobacco Use; Smoking Cessation | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a pragmatic, randomized, controlled, superiority trial with two parallel groups.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor conducting the 6-month telephone interview to ascertain smoking status is blinded to the participant's group assignment. The assessor has no access to the allocation data or the participant's interaction history with the Telegram bot. Participants are not explicitly informed of their group strategy but cannot be fully blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telegram Bot Intervention Group (Experimental): Participants receive standard care PLUS the 6-month behavioral intervention delivered via the Telegram chatbot.
  Interventions: Behavioral: Telegram-based Smoking Cessation Support
- Standard Care Control Group (Other): Participants receive standard care only. They are connected to the Telegram bot but only complete baseline and follow-up surveys without receiving any active smoking cessation content.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Behavioral: Telegram-based Smoking Cessation Support — A 6-month behavioral intervention delivered via a Telegram chatbot. The intervention includes personalized daily motivational messages, cognitive-behavioral techniques for craving management, access to an SOS/craving support button, weekly check-ins, and relapse prevention protocols. Content is tailored based on user responses to questionnaires (Fagerström Test, Importance/Confidence scales) and engagement metrics.
  Arms: Telegram Bot Intervention Group
Other: Standard Care (in control arm) — Routine physician advice to quit smoking provided upon hospital discharge. This represents the current standard of care in the participating clinical centers.
  Arms: Standard Care Control Group

SUMMARY:
This randomized controlled trial will evaluate whether a 6-month behavioral intervention delivered via Telegram messenger increases smoking cessation rates in patients after myocardial infarction (MI).

Adult smokers hospitalized with acute MI who regularly use Telegram will be randomly assigned to either:

* INTERVENTION GROUP: Standard care plus a 6-month Telegram chatbot program providing personalized motivational messages, cognitive-behavioral techniques for craving management, and relapse prevention support.
* CONTROL GROUP: Standard care (routine physician advice to quit smoking) plus basic surveys via Telegram without therapeutic content.

The primary outcome is 30-day point prevalence abstinence at 6 months, verified by blinded telephone interview with participant and corroborating report from a close relative. Secondary outcomes include changes in cigarette consumption, nicotine dependence, motivation, and intervention engagement metrics.

This study addresses the critical gap in smoking cessation support after hospital discharge and could provide evidence for a scalable digital health solution in cardiac secondary prevention.

DETAILED DESCRIPTION:
The TELEGRAM-MI trial is a multicenter, randomized, controlled, assessor-blinded superiority study testing a digital behavioral intervention for smoking cessation in post-myocardial infarction patients.

BACKGROUND: Smoking cessation is the most effective modifiable risk factor for reducing mortality after MI, yet long-term abstinence remains challenging due to limited sustained support. Digital interventions using popular messaging platforms offer a scalable solution to bridge the post-discharge support gap.

OBJECTIVES:

Primary: To determine if a 6-month Telegram chatbot intervention increases 30-day point prevalence abstinence rates at 6 months compared to standard care alone.

Secondary: To examine associations between baseline characteristics (nicotine dependence, motivation), engagement metrics, and cessation success; and to assess intervention acceptability.

METHODS: Approximately 142 participants will be recruited from inpatient cardiology departments. After providing informed consent, participants will be randomized 1:1 via the chatbot to either the intervention group (standard care plus 6-month behavioral support) or control group (standard care plus data collection only). The intervention incorporates evidence-based techniques including motivational messaging, cognitive-behavioral strategies, and relapse prevention protocols.

OUTCOMES: The primary outcome is biochemically unverified 30-day point prevalence abstinence at 6 months, assessed via blinded telephone interview with participant and relative verification. Secondary outcomes include various smoking behavior metrics collected through the chatbot platform.

ANALYSIS: Primary analysis will follow intention-to-treat principles, with missing data imputed as smoking. Statistical analyses will include chi-square tests for primary outcome and regression models for secondary outcomes.

POTENTIAL IMPACT: If effective, this intervention represents a readily implementable, low-cost strategy to enhance secondary prevention in cardiac patients.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Age 18 years or older.
* Hospitalization with a confirmed diagnosis of acute myocardial infarction (MI), including both ST-elevation MI (STEMI) and non-ST-elevation MI (NSTEMI).
* Current smoker at the time of index MI: self-reported smoking of at least one cigarette per day in the month prior to hospitalization.
* Regular user of the Telegram messenger application (app installed on a personal smartphone).
* Possession of a smartphone with internet access and a valid phone number.
* Ability and willingness to provide contact information for a close relative or cohabiting person who can verify smoking status at follow-up.

Exclusion Criteria:

* Smoking cessation more than 1 month prior to the index MI hospitalization.
* Physical or cognitive impairment that prevents the use of a smartphone (e.g., severe visual/hearing impairment, inability to read or respond to messages).
* Inability to read and understand the Russian language fluently.
* Comorbid condition with a life expectancy of less than 1 year.
* Active severe mental illness (e.g., psychosis, severe untreated depression) that would impede understanding of the protocol or adherence.
* Unwillingness or inability to provide contact details for a close relative for outcome verification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
30-day point prevalence abstinence (PPA) | 6 months
  Proportion of participants who report abstinence from smoking for the past 30 days or more, verified by both participant self-report AND corroborating report from a close relative or cohabiting person during a telephone interview conducted by a blinded assessor. A positive outcome is recorded ONLY if both sources confirm abstinence. Participants with missing data (e.g., lost to follow-up) will be considered smokers in the primary analysis (intention-to-treat).

SECONDARY OUTCOMES:
7-day point prevalence abstinence (7-day PPA) | 1 month and 3 months
  Proportion of participants who report abstinence from smoking for the past 7 days. Assessed via the Telegram bot.
Change in cigarette consumption | Baseline, 1 month, 3 months, and 6 months
  Change from baseline in the self-reported number of cigarettes smoked per day. Assessed via the Telegram bot.
Score on the Fagerström Test for Nicotine Dependence (FTND) | Baseline and 6 months
  Change in nicotine dependence measured by the FTND questionnaire (score range 0-10, higher scores indicate greater dependence). Assessed via the Telegram bot.
Motivation to quit (Importance and Confidence Scales) | Baseline and 6 months
  Scores on self-rated scales (0-10) for the importance of quitting and confidence in the ability to quit. Assessed via the Telegram bot.
Participant engagement with the Telegram bot | 6 months
  Composite measure of engagement (dose) including: proportion of completed weekly check-ins, proportion of opened messages, number of SOS/craving button uses, number of active weeks. Metrics are automatically logged by the bot.
Intervention acceptability and satisfaction | 6 months
  Total score on a custom acceptability and satisfaction questionnaire (5-12 items) completed by participants in the intervention group via the Telegram bot. Higher scores indicate higher satisfaction.
Time to first relapse | 6 months
  Number of days from randomization to the first self-reported relapse (lapse) event. Assessed via continuous monitoring through the bot's check-in system.

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Kuznetsov, MD, Principal Investigator — Ulyanovsk Regional Clinical Hospital; Dmitry Sergeev, PhD, Study Director — ITMO University; Artemiy Okhotin, MPH, Study Director — ITMO University
Locations (1):
- Ulyanovsk Regional Clinical Hospital, Ulyanovsk, Ulyanovsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial, after de-identification, will be shared. This includes demographic data, smoking history, questionnaire responses (Fagerström Test, Importance/Confidence scales), intervention engagement metrics, and primary/secondary outcome data.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 12 months after main results publication and ending 5 years after publication. Data will be available for this period.
Access Criteria: Data will be available to researchers who provide a methodologically sound research proposal approved by an independent review committee. Proposals should be directed to the corresponding author. Requestors will need to sign a data access agreement specifying the purpose of analysis, commitment to secure data handling, and agreement not to attempt re-identification of participants.

REFERENCES:
- [Result] Olano-Espinosa E, Avila-Tomas JF, Minue-Lorenzo C, Matilla-Pardo B, Serrano Serrano ME, Martinez-Suberviola FJ, Gil-Conesa M, Del Cura-Gonzalez I; Dejal@ Group. Effectiveness of a Conversational Chatbot (Dejal@bot) for the Adult Population to Quit Smoking: Pragmatic, Multicenter, Controlled, Randomized Clinical Trial in Primary Care. JMIR Mhealth Uhealth. 2022 Jun 27;10(6):e34273. doi: 10.2196/34273. PMID 35759328
- [Result] Bricker JB, Sullivan BM, Mull KE, Lavista-Ferres J, Santiago-Torres M. Efficacy of a conversational chatbot for cigarette smoking cessation: Protocol of the QuitBot full-scale randomized controlled trial. Contemp Clin Trials. 2024 Dec;147:107727. doi: 10.1016/j.cct.2024.107727. Epub 2024 Oct 28. PMID 39490766
- [Result] Hayrumyan V, Harutyunyan A, Harutyunyan T. Smoking cessation after myocardial infarction: Findings from a cross-sectional survey in Armenia. Tob Prev Cessat. 2023 Dec 11;9:36. doi: 10.18332/tpc/174359. eCollection 2023. PMID 38090104
- [Result] Gerber Y, Rosen LJ, Goldbourt U, Benyamini Y, Drory Y; Israel Study Group on First Acute Myocardial Infarction. Smoking status and long-term survival after first acute myocardial infarction a population-based cohort study. J Am Coll Cardiol. 2009 Dec 15;54(25):2382-7. doi: 10.1016/j.jacc.2009.09.020. PMID 20082928
- [Result] Leosdottir M, Warjerstam S, Michelsen HO, Schlyter M, Hag E, Wallert J, Larsson M. Improving smoking cessation after myocardial infarction by systematically implementing evidence-based treatment methods. Sci Rep. 2022 Jan 12;12(1):642. doi: 10.1038/s41598-021-04634-5. PMID 35022490
- [Result] Wilson K, Gibson N, Willan A, Cook D. Effect of smoking cessation on mortality after myocardial infarction: meta-analysis of cohort studies. Arch Intern Med. 2000 Apr 10;160(7):939-44. doi: 10.1001/archinte.160.7.939. PMID 10761958